CLINICAL TRIAL: NCT02568943
Title: An Open-label, Multi-center, Expanded Treatment Protocol of Oral Panobinostat in Combination With Bortezomib and Dexamethasone in Patients With Relapsed, and Relapsed and Refractory Multiple Myeloma
Brief Title: An Expanded Treatment Protocol of Panobinostat in Combination Therapy for Relapsed, and Relapsed and Refractory Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLBH589D2001X
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myelome, MM, expanded treatment, panobinostat, bortezomib, dexamethasone, relapsed, refractory, LBH589
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Panobinostat (PAN [LBH589]) is an orally administered pan-deacetylase inhibitor (DACi) belonging to a structurally novel class of compounds deregulating cell proliferation and survival mechanisms of cancer cells.
  Other Names: LBH589

SUMMARY:
The purpose of this study is to provide oral panobinostat (PAN) treatment to relapsed or relapsed and refractory multiple myeloma patients who are without satisfactory treatment alternatives prior to the commercial availability* and reimbursement of panobinostat during the regulatory approval process. This protocol will acquire additional safety data on the use of panobinostat in combination with bortezomib (BTZ) and dexamethasone (Dex) in patients with relapsed or relapsed and refractory multiple myeloma. In this protocol, PAN must be administered in the defined regimen in combination with both BTZ and DEX.

*(Note: throughout this protocol "commercially available" means local health authority approval and a functional method for reimbursement)

DETAILED DESCRIPTION:
This is an open-label, single arm, multi-center study of oral panobinostat administered in combination with bortezomib and dexamethasone in patients with relapsed, and relapsed and refractory multiple myeloma.

* Panobinostat will be administered in combination with bortezomib and dexamethasone over 2 weeks in each 21 day cycle; the third week will be without administration of any drug.
* Treatment phase 1 will consist of 8, 21 day cycles (24 weeks). Patients with clinical benefit at the end of cycle 8 as per investigator assessment may continue to receive study treatment in phase 2 for a maximum of an additional 24 weeks.
* Patients who have not achieved or maintained at least "no change" (EBMT response criterion) by 8 cycles must discontinue from study treatment
* The protocol will remain open in each participating country until drug is commercially available and reimbursable or until July 2017, whichever comes first (except in Norway where this protocol will end by March 2016).

Dosing schedule for treatment is detailed below:

Treatment Phase 1 (weeks 1-24 starting C1D1)

* PAN given three times per week (TIW), weeks 1 & 2 of each 3-week cycle (Cycle days 1,3,5,8,10, and 12)
* BTZ given twice a week (BIW) weeks 1 & 2 of each 3-week cycle (Cycle days 1,4,8, and 11)
* Dex given for 2 days twice a week (BIW), with BTZ on weeks 1 & 2 of each 3-week cycle (Cycle days 1,2,4,5,8,9,11, and 12)

Treatment Phase 2 (24 weeks starting C9D1)

* PAN given TIW, weeks 1 & 2 of each 3-week cycle (Cycle days 1,3,5,8,10, and 12)
* BTZ given once a week, weeks 1 & 2 of each 3 week cycle (Cycle days 1 and 8)
* Dex for 2 days once a week with BTZ, weeks 1 & 2 of each 3-week cycle (Cycle days 1,2,8, and 9)

ELIGIBILITY:
Inclusion Criteria:

- Written informed consent must be obtained prior to any screening procedures

Patients eligible for inclusion in this study have to meet all of the following criteria:

1. 1. Patient's age is ≥ 18 years at the time of signing informed consent
2. 2. Patient has a previous diagnosis of multiple myeloma, based on IMWG 2014 definitions. All three of the following criteria had been met:

   * Monoclonal immunoglobulin (M component) on electrophoresis, and on immunofixation on serum or on total 24 hour urine (or demonstration of M protein in cytoplasm of plasma cell for non-secretory myeloma).
   * Bone marrow (clonal) plasma cells ≥ 10% or biopsy proven plasmacytoma
   * Related organ or tissue impairment (CRAB symptoms: anemia, hypercalcemia, lytic bone lesions, renal insufficiency, hyperviscosity, amyloidosis or recurrent infections)
3. 3. Patient with multiple myeloma (Palumbo 2014) that is relapsed or relapsed and refractory to at least twoone prior lines of therapy and requires retreatment.

   1. Relapsed, defined by disease that recurred in a patient that responded under at least two prior therapiesy, by reaching a MR or better, and had not progressed under current therapy or up to 60 days of last dose of this therapy. Patients previously treated with bortezomib are eligible.
   2. Relapsed-and-refractory to a therapy, provided that patient meets both conditions:

      * patient has relapsed to at least twoone prior lines
      * and patient was refractory to at least twoone prior lines by either not reaching a MR, or progressed while under this therapy, or within 60 days of its last dose. Patients previously treated with bortezomib are eligible even if they are deemed refractory (based on results on Panorama 2)
   3. Patients who have previously received high dose therapy/autologous stem cell transplant are eligible.
   4. Patients who have undergone allogeneic stem cell transplant and do not have active graft vs host disease requiring immunosuppressive therapy are eligible.
4. 4. Patient has measurable disease at study screening defined by IMWG 2014 criteria (Palumbo 2014))
5. 5. A patient treated with local radiotherapy with or without concomitant exposure to steroids for pain control or management of cord/nerve root compression is eligible. Four weeks should have lapsed since last date of radiotherapy, which is recommended to be a limited field. Patients who require concurrent radiotherapy should have entry to the study deferred until the radiotherapy is completed and 2 weeks have passed since the last date of therapy.
6. 6. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
7. 7. Patient has the following laboratory values within 3 weeks before starting study drug (lab tests may be repeated, as clinically indicated, to obtain acceptable values before failure at screening is concluded but supportive therapies [such as erythropoietin and GCSF] are not to be administered within the week prior to screening tests for ANC or platelet count)

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109 /L
   2. Platelet count ≥ 100 x 109 /L
   3. Serum potassium, magnesium, phosphorus, within normal limits (WNL) for institution
   4. Total serum calcium (corrected for serum albumin) or ionized serum calcium greater than or equal to lower normal limits (> LLN) for institution, and not higher than CTCAE grade 1 in case of elevated value Note: Potassium, calcium, magnesium, and/or phosphorus supplements may be given to correct values that are < LLN.
   5. AST/SGOT and ALT/SGPT ≤ 2.5 x ULN
   6. Serum total bilirubin ≤ 1.5 x ULN (or ≤ 3.0 x ULN if patient has Gilbert syndrome)
   7. Serum creatinine levels ≤ 2.5 x ULN, or calculated creatinine clearance ≥ 30 ml/min
8. 8. Patient is able to swallow capsules
9. 9. Patient must be able to adhere to the study visit schedule and other protocol requirements
10. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at baseline

Exclusion Criteria:

-

Patients eligible for this study must not meet any of the following criteria:

1. 1. Patient has shown intolerance to bortezomib, dexamethasone or panobinostat or components of these drugs or has any contraindications to any of these therapies following locally applicable prescribing information.
2. 2. Patient is refractory to panobinostat
3. 3. Allogeneic stem cell transplant recipient presenting with graft versus host disease either active or requiring immunosuppression
4. 4. Patient has grade ≥ 2 peripheral neuropathy
5. 5. Patient taking any anti-cancer therapy concomitantly (bisphosphonates are permitted)
6. 6. Patient has second primary malignancy < 3 years of first dose of study treatment (except for adequately treated basal or squamous cell carcinoma, or in situ cancer of the cervix)
7. 7. Patient who received:

   1. Anti-myeloma chemotherapy or medication including IMiDs, proteasome inhibitor, and dexamethasone ≤3weeks prior to the start of study
   2. Experimental therapy or biologic immunotherapy including monoclonal antibodies ≤ 4 weeks prior to the start of study
   3. Prior radiation therapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to the start of study
8. 8. Patient has not recovered from all therapy-related toxicities associated with above listed treatments to < grade 2 CTCAE
9. 9. Patient has undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects to such therapy to < grade 2 CTCAE
10. 10. Patient with evidence of mucosal or internal bleeding
11. 11. Patient has unresolved diarrhea ≥ CTCAE grade 2
12. 12. Patient has impaired cardiac function, including any one of the following:

    1. History or presence of ventricular tachyarrhythmia
    2. Resting bradycardia defined as < 50 beats per minute
    3. QTcF > 450 msec on screening ECG
    4. Complete left bundle branch block (LBBB), bifascicular block
    5. Any clinically significant ST segment and/or T-wave abnormalities
    6. Presence of unstable atrial fibrillation (ventricular response rate > 100 bpm). Patients with stable atrial fibrillation can be enrolled provided they do not meet other cardiac exclusion criteria.
    7. Myocardial infarction or unstable angina pectoris ≤ 6 months prior to starting study drug
    8. Symptomatic congestive heart failure (New York Heart Association class III-IV)
    9. Other clinically significant heart disease and vascular disease (e.g. uncontrolled hypertension)
13. 13. Patient taking medications with relative risk or prolonging the QT interval or inducing Torsades de pointes, if such treatment cannot be discontinued or switched to a different medication prior to starting study drug
14. 14. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat (e.g. ulcerative disease, uncontrolled nausea, vomiting, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
15. 15. Patient has any other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease including dyspnea at rest from any cause, uncontrolled thyroid dysfunction) that could cause unacceptable safety risks or compromise compliance with the protocol
16. 16. Patient has a known history of HIV seropositivity (a test for screening is not required)
17. 17. Patient has active or chronic hepatitis B or C with or without evidence of hepatic insufficiency. However, patients who have received the hepatitis B vaccine or who have had hepatitis B and cleared the infection may be treated. Patients with hepatitis C who have undergone treatment with IFN and/or other antiviral agents can be considered for enrollment on a case by case basis after discussion with Novartis.
18. 18. Patient is a male not willing to use a barrier method of contraception (a condom) during the study and for 3 months after treatment with study drug has been completed.
19. 19. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
20. 20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after the final dose of study treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
    * Combination of any two of the following (a+b or a+c, or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- Austria (5):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Canada (3):
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Germany (25):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mutlangen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Winnenden
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Amman, Jordan
- Norway (2):
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Trondheim
- Sweden (3):
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå